CLINICAL TRIAL: NCT02500797
Title: Randomized Phase II Study of Nivolumab With or Without Ipilimumab in Patients With Metastatic or Unresectable Sarcoma
Brief Title: Nivolumab With or Without Ipilimumab in Treating Patients With Metastatic Sarcoma That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00260; NCI-2015-00260 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A091401; A091401 (Other: Alliance for Clinical Trials in Oncology); A091401 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Locally Advanced Bone Sarcoma; Locally Advanced Dedifferentiated Liposarcoma; Locally Advanced Gastrointestinal Stromal Tumor; Locally Advanced Soft Tissue Sarcoma; Metastatic Bone Sarcoma; Metastatic Liposarcoma; Metastatic Soft Tissue Sarcoma; Metastatic Undifferentiated Pleomorphic Sarcoma; Metastatic Unresectable Sarcoma; Pleomorphic Liposarcoma; Stage III Bone Sarcoma AJCC v7; Stage III Soft Tissue Sarcoma AJCC v7; Stage IV Bone Sarcoma AJCC v7; Stage IV Soft Tissue Sarcoma AJCC v7; Stage IVA Bone Sarcoma AJCC v7; Stage IVB Bone Sarcoma AJCC v7; Unresectable Bone Sarcoma; Unresectable Dedifferentiated Liposarcoma; Unresectable Liposarcoma; Unresectable Malignant Gastrointestinal Stromal Tumor; Unresectable Soft Tissue Sarcoma
MeSH Terms: conditions — Bone Neoplasms; Liposarcoma; Sarcoma; Histiocytoma, Malignant Fibrous | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (nivolumab) (Experimental): Patients receive nivolumab IV over 30 minutes once every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients who progress after 10 weeks on single agent nivolumab may elect to cross over to Arm II.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Quality-of-Life Assessment
- Arm II (nivolumab, ipilimumab) (Experimental): Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 90 minutes once every 3 weeks for 12 weeks. Patients then receive nivolumab IV over 30 minutes every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients who progress by imaging during the first 12 weeks of therapy may continue treatment, at the discretion of the patient and treating investigator.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm II (nivolumab, ipilimumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase II trial studies how well nivolumab with or without ipilimumab works in treating patients with sarcoma that has spread from the primary site to other parts of the body (metastatic) or cannot be removed by surgery (unresectable). Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. It is not yet known whether nivolumab works better with or without ipilimumab in treating patients with metastatic or unresectable sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the confirmed response rate of single agent nivolumab and dual agent nivolumab plus ipilimumab in patients with locally advanced/unresectable or metastatic soft tissue sarcoma.

SECONDARY OBJECTIVES:

I. To evaluate adverse event rates (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v]4.0) within each treatment arm.

II. To evaluate duration of response, clinical benefit rate, time to progression, progression-free survival, and overall survival within each treatment arm.

CORRELATIVE SCIENCE OBJECTIVES:

I. To potentially detect an early signal of confirmed response rate within a histologically defined patient cohort.

II. To assess the potential association between programmed cell death 1 ligand 1 (PD-L1) expression (by immunohistochemistry [IHC]) and clinical outcome, within each treatment.

III. To evaluate associations between selected biomarker measured in serial peripheral blood and with clinical efficacy, within each treatment.

IV. To evaluate the association between selected biomarker measured in tumor tissue with clinical efficacy, within each treatment.

V. To evaluate the association between baseline tumor mutational burden and neoantigen production with clinical efficacy within each treatment.

EXPLORATORY PHASE II OBJECTIVES (CROSSOVER TREATMENT):

I. To evaluate secondary endpoints within patients crossing over to dual agent nivolumab plus ipilimumab after experiencing progressive disease while receiving single agent nivolumab.

II. To evaluate correlative science objectives endpoints within patients crossing over to dual agent nivolumab plus ipilimumab after experiencing progressive disease while receiving single agent nivolumab.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive nivolumab intravenously (IV) over 30 minutes once every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients who progress after 10 weeks on single agent nivolumab may elect to cross over to Arm II.

ARM II: Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 90 minutes once every 3 weeks for 12 weeks. Patients then receive nivolumab IV over 30 minutes every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients who progress by imaging during the first 12 weeks of therapy may continue treatment, at the discretion of the patient and treating investigator.

After completion of study treatment, patients are followed up at 4 weeks and then every 6 months 3 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION ELIGIBILITY CRITERIA:
* Patients must have a formalin-fixed, paraffin-embedded (FFPE) tumor block OR 1 representative hematoxylin and eosin (H&E) and 20 unstained sarcoma tissue slides available for submission to central pathology review; this review is mandatory prior to registration to confirm eligibility
* REGISTRATION ELIGIBILITY CRITERIA:
* Patients must have histologically confirmed bone or soft tissue sarcoma by central pathology review

  * Patients must have histologically confirmed liposarcoma (LPS) (only dedifferentiated and pleomorphic; well differentiated not eligible), undifferentiated pleomorphic sarcoma (UPS)/malignant fibrous histiocytoma (MFH), or gastrointestinal stromal tumor (GIST)
* Measurable disease
* Locally advanced/unresectable or metastatic disease
* >= 1 prior systemic therapy for sarcoma, including adjuvant systemic therapy
* No prior therapy with ipilimumab or nivolumab, or any agent targeting programmed cell death 1 (PD-1), PD-L1 or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4)
* No treatment with biologic therapy, immunotherapy, chemotherapy, investigational agent for malignancy, or radiation =< 28 days before study registration; no treatment with nitrosourea or mitomycin =< 42 days before study registration; for GIST, tyrosine kinase inhibitor can be continued for up to 3 days prior to initiation of study treatment
* Patients should have resolution of any toxic effects of prior therapy (except alopecia) to NCI CTCAE, version 4.0, grade 1 or less
* No history of the following:

  * Active known or suspected autoimmune disease
  * Patients with human immunodeficiency virus (HIV) are eligible if the lymphocytes > 350 cluster of differentiation (CD)4+ cells and no detectable viral load
  * Symptomatic, untreated, or uncontrolled brain metastases present
  * Active autoimmune colitis
  * Autoimmune panhypopituitarism
  * Autoimmune adrenal insufficiency
  * Known active hepatitis B or C

    * Hepatitis B can be defined as:

      * Hepatitis B surface antigen (HBsAg) > 6 months
      * Serum hepatitis B virus (HBV) deoxyribonucleic acid (DNA) 20,000 IU/ml (105 copies/ml), lower values 2,000-20,000 IU/ml (104-105 copies/ml) are often seen in hepatitis B e antigen (HBeAg)-negative chronic hepatitis B
      * Persistent or intermittent elevation in alanine aminotransferase (ALT)/alanine aminotransferase (AST) levels
      * Liver biopsy showing chronic hepatitis with moderate or severe necroinflammation
    * Hepatitis C can be defined as:

      * Hepatitis C antibody (Ab) positive
      * Presence of hepatitis C virus (HCV) ribonucleic acid (RNA)
  * Known active pulmonary disease with hypoxia defined as:

    * Oxygen saturation < 85% on room air or
    * Oxygen saturation < 88% despite supplemental oxygen
* No systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of registration
* Not pregnant and not nursing because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects; therefore for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine =< 1.5 x upper limit of normal (ULN) OR calculated (calc.) creatinine clearance > 45 mL/min using the lean body mass formula only (Modified Cockcroft and Gault; Shargel and Yu 1985)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) in absence of Gilbert disease (total bilirubin =< 3 x ULN with Gilbert); also, if hyperbilirubinemia is clearly attributed to liver metastases total bilirubin =< 3 x ULN is permitted
* AST/ALT =< 3 x upper limit of normal (ULN)
* Thyroid stimulating hormone (TSH) within normal limits (WNL); supplementation is acceptable to achieve a TSH WNL; in patients with abnormal TSH if free T4 is normal and patient is clinically euthyroid, patient is eligible
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): Measurable disease
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): Locally advanced/unresectable or metastatic disease
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): Patient MUST have had progressive disease (radiographic or clinical) while on arm 1 single agent nivolumab while registered to A091401
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): Patients removed from any immunotherapy for reasons other than progressive disease, including arm 1 single agent nivolumab of A091401, are NOT eligible for re-registration
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): Patients must have completed a minimum of 10 weeks of single agent nivolumab on arm 1 of A091401 to be eligible for re-registration
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): Patients must have completed study drug on arm 1 of A091401 (i.e., last dose of nivolumab) =< 12 months of re-registration to crossover dual agent therapy
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): No treatment with immunotherapy =< 21 days before re-registration; no treatment with biologic therapy, chemotherapy, investigational agent for malignancy, or radiation =< 28 days before re-registration; no treatment with nitrosourea or mitomycin =< 42 days before re-registration
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): Patients should have resolution of any toxic effects of prior therapy (except fatigue and alopecia) to NCI CTCAE, version 4.0, grade 1 or less, including immune toxicity
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): No systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of re-registration
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): Not pregnant and not nursing because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects; therefore, for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to re-registration is required
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): ECOG performance status 0 or 1
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): ANC >= 1,500/mm^3
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): Platelet count >= 100,000/mm^3
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): Creatinine =< 1.5 ULN OR calc. creatinine clearance > 45 mL/min (using lean body mass formula only [Modified Cockcroft and Gault; Shargel and Yu 1985])
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): Total bilirubin =< 1.5 x ULN in absence of Gilbert disease (total bilirubin =< 3 x ULN with Gilbert); if hyperbilirubinemia is clearly attributed to liver metastases, total bilirubin =< 3 x ULN is permitted
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): AST/ALT =< 3 x ULN
* RE-REGISTRATION ELIGIBILITY CRITERIA (FOR PATIENTS WHO CROSSOVER FROM ARM 1 NIVOLUMAB ALONE TO DUAL AGENT NIVOLUMAB AND IPILIMUMAB UPON PROGRESSION): TSH WNL; supplementation is acceptable to achieve a TSH WNL; in patients with abnormal TSH, if free T4 is normal and patient is clinically euthyroid, patient is eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra P D'Angelo, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (651):
- United States (651):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - Sutter Davis Hospital, Davis, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - William Beaumont Hospital-Grosse Pointe, Grosse Pointe, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon Rectal Associates, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Hematology Oncology Consultants PC, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Ocean University Medical Center, Brick, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Bayshore Community Hospital, Holmdel, New Jersey
  - Southern Ocean County Medical Center, Manahawkin, New Jersey
  - Cooper CyberKnife Center, Mount Laurel, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Glens Falls Hospital, Glens Falls, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Seligson ND, Chen JL, Goodrich AC, Van Tine BA, Campbell JD, Richards AL, Antonescu CR, Liebner DA, Milhem MM, Streicher H, Tap WD, Schwartz GK, George S, D'Angelo SP. A multicenter, randomized, non-comparative, phase II study of nivolumab +/- ipilimumab for patients with metastatic sarcoma (Alliance A091401): expansion cohorts and correlative analyses. J Immunother Cancer. 2024 Sep 28;12(9):e009472. doi: 10.1136/jitc-2024-009472. PMID 39343511
- [Derived] D'Angelo SP, Mahoney MR, Van Tine BA, Atkins J, Milhem MM, Jahagirdar BN, Antonescu CR, Horvath E, Tap WD, Schwartz GK, Streicher H. Nivolumab with or without ipilimumab treatment for metastatic sarcoma (Alliance A091401): two open-label, non-comparative, randomised, phase 2 trials. Lancet Oncol. 2018 Mar;19(3):416-426. doi: 10.1016/S1470-2045(18)30006-8. Epub 2018 Jan 19. PMID 29370992

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: GIST Cohort: 24 patients assessed for eligibility; 3 excluded (i.e. ineligible) and 21 randomized.> LPS Cohort: 37 patients assessed for eligibility; 11 excluded, 3 included (2 pre-registered as UPS/MFH cohort, 1 pre-registered as GIST cohort) and 29 randomized.> UPS/MFH Cohort: 47 patients assessed for eligibility; 18 excluded and 29 randomized.
Groups:
- Initial Cohort - Arm I (Nivolumab): Patients receive 3mg/kg nivolumab IV over 30 minutes once every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients who progress on single agent nivolumab may elect to cross over to Initial Cohort - Arm II.
- Initial Cohort - Arm II (Nivolumab, Ipilimumab): Patients receive 3mg/kg nivolumab IV over 30 minutes and 1mg/kg ipilimumab IV over 90 minutes once every 3 weeks for 12 weeks. Patients then receive 3mg/kg nivolumab IV over 30 minutes every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity.
- Expansion LPS Cohort - Arm I (Nivolumab): Dedifferentiated liposarcoma (LPS) Cohort Patients receive 3mg/kg nivolumab IV over 30 minutes once every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients who progress after 10 weeks on single agent nivolumab may elect to cross over to LPS Cohort - Arm II.
- Expansion LPS Cohort - Arm II (Nivolumab, Ipilimumab): Dedifferentiated liposarcoma (LPS) Cohort Patients receive 3mg/kg nivolumab IV over 30 minutes and 1mg/kg ipilimumab IV over 90 minutes once every 3 weeks for 12 weeks. Patients then receive 3mg/kg nivolumab IV over 30 minutes every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients who progress by imaging during the first 12 weeks of therapy may continue treatment, at the discretion of the patient and treating investigator.
- Expansion UPS/MFH Cohort - Arm I (Nivolumab): Undifferentiated Pleomorphic Sarcoma & Malignant Fibrous Histiocytoma (UPS/MFH) Cohort Patients receive 3mg/kg nivolumab IV over 30 minutes once every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients who progress after 10 weeks on single agent nivolumab may elect to cross over to UPS/MFH Cohort - Arm II.
- Expansion UPS/MFH Cohort - Arm II (Nivolumab, Ipilimumab): Undifferentiated Pleomorphic Sarcoma & Malignant Fibrous Histiocytoma (UPS/MFH) Cohort Patients receive 3mg/kg nivolumab IV over 30 minutes and 1mg/kg ipilimumab IV over 90 minutes once every 3 weeks for 12 weeks. Patients then receive 3mg/kg nivolumab IV over 30 minutes every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients who progress by imaging during the first 12 weeks of therapy may continue treatment, at the discretion of the patient and treating investigator.
- Expansion GIST Cohort - Arm I (Nivolumab): Gastrointestinal stromal tumor (GIST) Cohort Patients receive 3mg/kg nivolumab IV over 30 minutes once every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients who progress after 10 weeks on single agent nivolumab may elect to cross over to GIST Cohort - Arm II.
- Expansion GIST Cohort - Arm II (Nivolumab, Ipilimumab): Gastrointestinal stromal tumor (GIST) Cohort Patients receive 3mg/kg nivolumab IV over 30 minutes and 1mg/kg ipilimumab IV over 90 minutes once every 3 weeks for 12 weeks. Patients then receive 3mg/kg nivolumab IV over 30 minutes every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients who progress by imaging during the first 12 weeks of therapy may continue treatment, at the discretion of the patient and treating investigator.
Period: Overall Study
Arm/Group | Initial Cohort - Arm I (Nivolumab) | Initial Cohort - Arm II (Nivolumab, Ipilimumab) | Expansion LPS Cohort - Arm I (Nivolumab) | Expansion LPS Cohort - Arm II (Nivolumab, Ipilimumab) | Expansion UPS/MFH Cohort - Arm I (Nivolumab) | Expansion UPS/MFH Cohort - Arm II (Nivolumab, Ipilimumab) | Expansion GIST Cohort - Arm I (Nivolumab) | Expansion GIST Cohort - Arm II (Nivolumab, Ipilimumab)
Started | 43 | 42 | 15 | 14 | 14 | 15 | 10 | 11
Arm I Crossover (Arm I Patients who progress after 10 weeks on single agent nivolumab and cross over to Arm II.) | 4 | 0 | 6 | 0 | 1 | 0 | 2 | 0
Completed | 42 | 42 | 15 | 14 | 13 | 14 | 10 | 11
Not Completed | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Cancel (rapid disease progression) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized patients are included in this analysis.
Groups:
- Initial Single: Patients receive 3mg/kg nivolumab IV over 30 minutes once every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity.
- Initial Dual: Patients receive 3mg/kg nivolumab IV over 30 minutes and 1mg/kg ipilimumab IV over 90 minutes once every 3 weeks for 12 weeks. Patients then receive 3mg/kg nivolumab IV over 30 minutes every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity.
- LPS Single: Dedifferentiated liposarcoma (LPS) Cohort Patients receive 3mg/kg nivolumab IV over 30 minutes once every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity.
- LPS Dual: Dedifferentiated liposarcoma (LPS) Cohort Patients receive 3mg/kg nivolumab IV over 30 minutes and 1mg/kg ipilimumab IV over 90 minutes once every 3 weeks for 12 weeks. Patients then receive 3mg/kg nivolumab IV over 30 minutes every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients who progress by imaging during the first 12 weeks of therapy may continue treatment, at the discretion of the patient and treating investigator.
- UPS/MFH Single: Undifferentiated Pleomorphic Sarcoma & Malignant Fibrous Histiocytoma (UPS/MFH) Cohort Patients receive 3mg/kg nivolumab IV over 30 minutes once every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity.
- UPS/MFH Dual: Undifferentiated Pleomorphic Sarcoma & Malignant Fibrous Histiocytoma (UPS/MFH) Cohort Patients receive 3mg/kg nivolumab IV over 30 minutes and 1mg/kg ipilimumab IV over 90 minutes once every 3 weeks for 12 weeks. Patients then receive 3mg/kg nivolumab IV over 30 minutes every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients who progress by imaging during the first 12 weeks of therapy may continue treatment, at the discretion of the patient and treating investigator.
- GIST Single: Gastrointestinal stromal tumor (GIST) Cohort Patients receive 3mg/kg nivolumab IV over 30 minutes once every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity.
- GIST Dual: Gastrointestinal stromal tumor (GIST) Cohort Patients receive 3mg/kg nivolumab IV over 30 minutes and 1mg/kg ipilimumab IV over 90 minutes once every 3 weeks for 12 weeks. Patients then receive 3mg/kg nivolumab IV over 30 minutes every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients who progress by imaging during the first 12 weeks of therapy may continue treatment, at the discretion of the patient and treating investigator.
- Total: Total of all reporting groups
Arm/Group | Initial Single | Initial Dual | LPS Single | LPS Dual | UPS/MFH Single | UPS/MFH Dual | GIST Single | GIST Dual | Total
Number analyzed (Participants) | 43 | 42 | 15 | 14 | 14 | 15 | 10 | 11 | 164
Age, Continuous [Median (Full Range); unit: years] | 56.0 [21.0 to 76.0] | 57.0 [27.0 to 81.0] | 62.0 [27.0 to 82.0] | 58.5 [46.0 to 68.0] | 63.5 [34.0 to 85.0] | 60.0 [44.0 to 84.0] | 69.0 [41.0 to 79.0] | 62.0 [40.0 to 81.0] | 62 [27 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 8 | 5 | 5 | 8 | 2 | 5 | 77
  Male | 22 | 19 | 7 | 9 | 9 | 7 | 8 | 6 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Black or African American | 4 | 3 | 0 | 0 | 2 | 1 | 2 | 0 | 12
  White | 38 | 34 | 15 | 13 | 12 | 13 | 7 | 10 | 142
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 5
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 28 | 24 | 6 | 8 | 3 | 7 | 6 | 8 | 90
    1 | 15 | 18 | 9 | 6 | 11 | 8 | 4 | 3 | 74

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a Confirmed Response
Description: The number of participants who achieved a confirmed response is defined as the number of patients having a best objective tumor status of complete response (CR) or partial response (PR) lasting at least 4 weeks as determined using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. (CR: Disappearance of all evidence of disease, PR: Regression of measurable disease and no new sites).
Time Frame: Up to 44 months
Population: Participants who completed the study and were evaluable for the primary endpoint are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Single | Initial Dual | LPS Single | LPS Dual | UPS/MFH Single | UPS/MFH Dual | GIST Single | GIST Dual
Number analyzed (Participants) | 42 | 42 | 15 | 14 | 13 | 14 | 10 | 11
Participants | 2 | 6 | 1 | 2 | 1 | 2 | 0 | 0

2. Secondary Outcome: Number of Participants Who Experienced at Least One Grade 3 or Higher Adverse Event Regardless of Attribution
Description: The number of participants who experienced at least one grade 3 or higher adverse event (AE) regardless of attribution. AEs are graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (version 5.0 beginning April 1, 2018).
Time Frame: Up to 4 weeks after completion of study treatment
Population: Randomized patients who received treatment (i.e. exclude cancel patients).
Measure: Count of Participants; unit: Participants
Groups:
- Initial Single: Patients receive 3mg/kg nivolumab IV over 30 minutes once every 2 weeks. Cycles repeat every 42 days for up to 108 weeks in the absence of disease progression or unacceptable toxicity. Patients who progress on single agent nivolumab may elect to cross over to Initial Cohort - Arm II.
Arm/Group | Initial Single | Initial Dual | LPS Single | LPS Dual | UPS/MFH Single | UPS/MFH Dual | GIST Single | GIST Dual
Number analyzed (Participants) | 42 | 42 | 15 | 14 | 13 | 14 | 10 | 11
Participants
  Grade 3 Event | 19 | 25 | 11 | 5 | 9 | 6 | 5 | 6
  Grade 4 Event | 3 | 4 | 0 | 0 | 1 | 2 | 1 | 1
  Grade 5 Event | 5 | 6 | 1 | 0 | 3 | 1 | 1 | 0

3. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients who have achieved a confirmed response as the date at which the patient's objective status is first noted to be a CR or PR to the earliest date progression (PD) is documented. The distribution of duration of response will be estimated using the method of Kaplan-Meier. (CR: Disappearance of all evidence of disease, PR: Regression of measurable disease and no new sites, PD: Any new lesion or increase by >= 50% of previously involved sites from nadir).
Time Frame: Time from first response to progression, assessed up to 3 years
Population: Participants who achieved a confirmed response are included in this analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Initial Single | Initial Dual | LPS Single | LPS Dual | UPS/MFH Single | UPS/MFH Dual | GIST Single | GIST Dual
Number analyzed (Participants) | 2 | 6 | 1 | 2 | 1 | 2 | 0 | 0
months | 7.4 [3.2 to 11.6] | 6.2 [1.4 to 14.1] | 14.5 [14.5 to 14.5] | 10.675 [8.25 to 13.1] | 14.6 [14.6 to 14.6] | 3.19 [1.61 to 7.59] |  |

4. Secondary Outcome: 6-Month Clinical Benefit Rate [Initial Cohort]
Description: The 6-month clinical benefit rate is defined as the percentage of participants with a response or stable disease (CR, PR, or SD) at 6 months. (CR: Disappearance of all evidence of disease, PR: Regression of measurable disease and no new sites, PD: Any new lesion or increase by >= 50% of previously involved sites from nadir, SD: Not CR/PR or PD).
Time Frame: At 6 months
Population: Randomized Initial Cohort participants who received treatment (i.e. exclude cancel patients) Only.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Initial Single | Initial Dual
Number analyzed (Participants) | 42 | 42
percentage of participants | 10 [3 to 22] | 12 [6 to 28]

5. Secondary Outcome: 6-Month Clinical Benefit Rate [Expansion LPS and UPS/MFH Cohorts Only]
Description: as for outcome 4
Time Frame: At 6 months
Population: Randomized Expansion LPS and UPS/MFH Cohorts Participants who received treatment Only
Measure: Number (85% Confidence Interval); unit: percentage of participants
Arm/Group | LPS Single | LPS Dual | UPS/MFH Single | UPS/MFH Dual
Number analyzed (Participants) | 15 | 14 | 13 | 14
percentage of participants | 6.7 [NA to 21] — 1-sided Upper Confidence Limit | 35.7 [NA to 53.1] — 1-sided Upper Confidence Limit | 15.4 [NA to 32.7] — 1-sided Upper Confidence Limit | 35.7 [NA to 53.1] — 1-sided Upper Confidence Limit

6. Secondary Outcome: 6-Month Clinical Benefit Rate [Expansion GIST Cohort Only]
Description: as for outcome 4
Time Frame: At 6 months
Population: Randomized Expansion GIST Cohort Participants who received treatment Only.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | GIST Single | GIST Dual
Number analyzed (Participants) | 10 | 11
percentage of participants | 10 [NA to 27.1] — 1-sided Upper Confidence Limit | 54.5 [NA to 70.1] — 1-sided Upper Confidence Limit

7. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression (PD) is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator. (PD: Any new lesion or increase by >= 50% of previously involved sites from nadir).
Time Frame: Time from randomization to first of either disease progression or death from any cause, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Initial Single | Initial Dual | LPS Single | LPS Dual | UPS/MFH Single | UPS/MFH Dual | GIST Single | GIST Dual
Number analyzed (Participants) | 42 | 41 | 15 | 14 | 13 | 14 | 10 | 11
months | 1.7 [1.4 to 4.3] | 4.1 [2.6 to 4.7] | 4.6 [3.2 to NA] — The 95% Confidence Interval upper limit was not estimable (i.e. below the level of detection). | 5.5 [2.8 to NA] — The 95% Confidence Interval upper limit was not estimable (i.e. below the level of detection). | 1.5 [1.4 to NA] — The 95% Confidence Interval upper limit was not estimable (i.e. below the level of detection). | 2.7 [1.5 to NA] — The 95% Confidence Interval upper limit was not estimable (i.e. below the level of detection). | 1.5 [1.3 to 10] | 2.9 [1.4 to NA] — The 95% Confidence Interval upper limit was not estimable (i.e. below the level of detection).

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival time is defined as the time from randomization to death due to any cause. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Time from randomization to death from any cause, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Initial Single | Initial Dual | LPS Single | LPS Dual | UPS/MFH Single | UPS/MFH Dual | GIST Single | GIST Dual
Number analyzed (Participants) | 42 | 41 | 15 | 14 | 13 | 14 | 10 | 11
months | 10.7 [5.5 to 15.4] | 14.3 [9.6 to NA] — The 95% Confidence Interval Upper Limit was not estimable (i.e. below the level of detection.) | 8.1 [7 to NA] — The 95% Confidence Interval Upper Limit was not estimable (i.e. below the level of detection.) | 13.1 [9.1 to NA] — The 95% Confidence Interval Upper Limit was not estimable (i.e. below the level of detection.) | 6.6 [2.4 to 17.6] | NA [NA to NA] — The median has not yet been reached and the 95% Confidence Interval was not estimable. | 9.1 [4.9 to NA] — The 95% Confidence Interval Upper Limit was not estimable (i.e. below the level of detection.) | 12.2 [6 to NA] — The 95% Confidence Interval Upper Limit was not estimable (i.e. below the level of detection.)

9. Other Pre Specified Outcome: PD-L1 Expression Assessed Using Immunohistochemistry (IHC)
Description: Categorical data analysis and logistic regression will be used to evaluate the associations between PD-L1 expression (by IHC) and clinical outcome (e.g., response, clinical benefit, progression-free survival, and survival). Kaplan-Meier methodology and Cox proportional hazards models will be used to evaluate time to event endpoints.
Time Frame: Up to 3 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Selected Biomarkers Measured in Serial Peripheral Blood
Description: Summary statistics will be used to for describing changes across time. The time course of biomarker outcomes will be investigated graphically, by summary plots or individual patient plots. If there is suggestion of meaningful trend, methods such as linear mixed models may be used to characterize the pattern of change over time. Kaplan-Meier methodology and Cox proportional hazards models will be used to evaluate time to event endpoints.
Time Frame: Baseline to up to 3 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Selected Biomarkers Measured in Tumor Tissue
Description: Categorical data analysis and logistic regression will be used to correlated biomarkers with and clinical outcome (e.g., response, clinical benefit, time to progression, progression free survival, and survival) within each study component. Kaplan-Meier methodology and Cox proportional hazards models will be used to evaluate time to event endpoints.
Time Frame: Up to week 6
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Confirmed Response in Patients Who Crossover From Single Agent Nivolumab to Dual Agent Treatment Following Progression
Description: Confirmed response will be evaluated in patients who crossover from single agent nivolumab to dual agent treatment following progression.
Time Frame: Up to 3 years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Duration of Response in Patients Who Crossover From Single Agent Nivolumab to Dual Agent Treatment Following Progression
Description: Evaluated using Kaplan-Meier methodology.
Time Frame: Time from first response to progression, assessed up to 3 years
Reporting Status: Not Posted

14. Other Pre Specified Outcome: PFS in Patients Who Crossover From Single Agent Nivolumab to Dual Agent Treatment Following Progression
Description: Evaluated using Kaplan-Meier methodology.
Time Frame: Time from randomization to first of either disease progression or death from any cause, assessed up to 3 years
Reporting Status: Not Posted

15. Other Pre Specified Outcome: OS in Patients Who Crossover From Single Agent Nivolumab to Dual Agent Treatment Following Progression
Description: Evaluated using Kaplan-Meier methodology.
Time Frame: Time from randomization to death from any cause, assessed up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 4 weeks after completion of study treatment; up to 44 months
Description: Serious AEs and Other (Not Including Serious) AEs summary tables summarizes AEs assessed for participants who started treatment and were evaluable for AEs. All-cause mortality is assessed for all enrolled participants. Adverse events are described and graded using the terminology and grading categories defined in the NCI's Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0. However, CTCAE v5.0 is used for serious AE reporting through CTEP-AERS as of April 1, 2018.
Arm/Group | Initial Single | Initial Dual | LPS Single | LPS Dual | UPS/MFH Single | UPS/MFH Dual | GIST Single | GIST Dual
All-Cause Mortality (participants affected / at risk) | 37/43 | 34/42 | 11/15 | 10/14 | 10/14 | 7/15 | 8/10 | 7/11
Serious Adverse Events (participants affected / at risk) | 19/42 | 21/42 | 9/15 | 1/14 | 8/13 | 7/14 | 5/10 | 6/11
Other Adverse Events (participants affected / at risk) | 39/42 | 40/42 | 15/15 | 14/14 | 12/13 | 14/14 | 10/10 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Single (N=42) | Initial Dual (N=42) | LPS Single (N=15) | LPS Dual (N=14) | UPS/MFH Single (N=13) | UPS/MFH Dual (N=14) | GIST Single (N=10) | GIST Dual (N=11)
Anemia (Blood and lymphatic system disorders) | 4 (5) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papilledema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jejunal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intraoperative urinary injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Single (N=42) | Initial Dual (N=42) | LPS Single (N=15) | LPS Dual (N=14) | UPS/MFH Single (N=13) | UPS/MFH Dual (N=14) | GIST Single (N=10) | GIST Dual (N=11)
Anemia (Blood and lymphatic system disorders) | 10 (13) | 10 (16) | 3 (5) | 3 (6) | 2 (3) | 3 (7) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 6 (10) | 7 (28) | 3 (6) | 2 (4) | 1 (1) | 4 (14) | 1 (9) | 2 (8)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 11 (21) | 11 (19) | 9 (20) | 8 (18) | 1 (2) | 1 (7) | 7 (9) | 8 (22)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (8) | 6 (13) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (6) | 13 (15) | 6 (13) | 6 (9) | 3 (4) | 5 (5) | 2 (4) | 6 (15)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (17) | 12 (18) | 7 (12) | 5 (11) | 2 (4) | 5 (10) | 3 (10) | 6 (9)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 2 (7)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 27 (58) | 29 (71) | 12 (27) | 13 (43) | 9 (14) | 11 (32) | 9 (14) | 6 (23)
Fever (General disorders) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 3 (6) | 2 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gum infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (5) | 3 (3) | 0 (0) | 2 (2) | 1 (2) | 3 (4) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (4) | 3 (4) | 2 (2) | 4 (7) | 0 (0) | 1 (2) | 1 (7) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 1 (2) | 4 (5) | 2 (9) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 3 (8) | 2 (3)
Creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
GGT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 3 (3) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Lymphocyte count decreased (Investigations) | 5 (7) | 3 (3) | 4 (10) | 1 (2) | 1 (1) | 2 (2) | 1 (3) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 1 (2) | 1 (3) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (6) | 1 (3) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 12 (18) | 14 (21) | 10 (20) | 3 (4) | 5 (7) | 7 (8) | 5 (7) | 5 (11)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (10) | 3 (4) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4) | 3 (4) | 3 (4) | 2 (2) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 2 (3) | 4 (6) | 1 (2) | 1 (1) | 3 (3) | 1 (2) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (16) | 8 (17) | 3 (5) | 6 (18) | 9 (12) | 6 (15) | 5 (5) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 8 (24) | 7 (11) | 6 (13) | 7 (10) | 5 (9) | 3 (7) | 3 (15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (19) | 10 (17) | 4 (5) | 3 (4) | 8 (14) | 2 (5) | 4 (6) | 3 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 2 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) | 3 (7) | 3 (10) | 4 (17) | 0 (0) | 1 (2) | 2 (14)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (7) | 4 (5) | 2 (5) | 2 (4) | 2 (3) | 1 (1) | 2 (4) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 2 (10) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 3 (6) | 1 (2) | 2 (2) | 0 (0) | 1 (6) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphedema (Vascular disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT02500797/Prot_SAP_000.pdf